CLINICAL TRIAL: NCT05984706
Title: What Difficulties Do Children and Adolescents Experience in Everyday Activities After a Traumatic Event? Focus Groups and Delphi Survey for the Development of a Questionnaire on PTSD-related Functional Impairment
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Principal Investigator, Lasse Bartels, Principal investigator, University Children's Hospital, Zurich
Other Study IDs: 2023-01290
Record Dates: First submitted 2023-07-21; First posted 2023-08-09 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-12

CONDITIONS: PTSD; Functioning, Psychosocial
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Trauma-exposed children and adolescents: Focus group and Delphi survey
  Interventions: Other: Focus groups and Delphi Questionnaire
- Caregivers of trauma-exposed children and adolescents: Focus group and Delphi survey
  Interventions: Other: Focus groups and Delphi Questionnaire
- Clinical experts: Delphi survey
  Interventions: Other: Focus groups and Delphi Questionnaire

INTERVENTIONS:
Other: Focus groups and Delphi Questionnaire — 1. Focus groups to identify relevant domains of PTSD-related functional impairment in trauma-exposed children and adolescents to ensure content validity. 2. Delphi Questionnaire evaluation of a list of domains of PTSD-related functional impairment in trauma-exposed children and adolescents (previously selected from based on a literature review and focus groups) on a Likert scale of 1 to 5 for their relevance

SUMMARY:
Post-traumatic Stress Disorder (PTSD) in children and adolescents is often associated with a myriad of significant impairments in daily functioning, including family relationships, school/work, leisure time activities, and social relationships. While a majority of attention has been placed on definition and assessment of post-traumatic stress symptoms (PTSS), less emphasis has been placed on the effect of PTSS on related functional impairment in daily life. The current assessment of PTSD-related functional impairment is conducted either with additional items inserted in PTSD measures that inquire about daily functioning or with the utilization of global functional impairment measures. The former approach is usually based on face validity only and varies content-wise. The latter approach often consists of scales that conflate symptoms with functioning, focus on impairment due to physical rather than mental health problems, and are not validated in trauma-exposed children and adolescents. Furthermore, scales usually do not include sufficient age-specific adjustments for younger children. Thus, the current assessment of PTSD-related functional impairment in children and adolescents demonstrates noteworthy shortcomings. Despite the well-recognized debilitating effect of PTSD on daily functioning, no measure has yet been developed to assess PTSD-related functional impairment tailored to trauma-exposed children and adolescents based on the input from the target population and their caregivers. The aim of this project is therefore to develop an instrument that assesses PTSD-related functional impairment in trauma-exposed children and adolescents (young children age 1-6 years (caregiver-report) as well as for older children and adolescents age 7-18 years (self- and caregiver-report)) by conducting focus groups and a Delphi survey.

ELIGIBILITY:
Inclusion Criteria:

The same inclusion criteria apply for the focus group discussions and for the Delphi process.

For children and adolescents:

* Children and adolescents, who experienced at least one PTE according to the DSM-5 definition of a traumatic event.
* The PTE(s) must have occurred after the fourth birthday.
* The PTE(s) must have occurred at least 1 month ago.
* Children and adolescents must be 7-18 years of age.
* Children and adolescents are either in trauma-focused treatment at the time of recruitment or they present with at least a moderate PTSS severity according to the Child and Adolescents Trauma Screen 2 (CATS-2) Self-report.
* Children and adolescents must have sufficient command of the German language, excluding a small group of 4-5 unaccompanied refugee adolescents who will also be included. This group will be assisted by an interpreter.
* The children and adolescents do not have any physical impairment due to injuries or somatic illnesses (self-assessment).
* The children and adolescents are not acute suicidal. The responsible psychotherapists or supervisors of the "Schlupfhuus" will provide information about it.

For caregivers:

* Caregivers of children and adolescents, who experienced at least one PTE according to the DSM-5 definition of a traumatic event.
* The PTE(s) must have occurred at least 1 month ago.
* The child or adolescent must be between 1-18 years of age.
* Children and adolescents are either in trauma-focused therapy at the time of recruitment or they present with at least a moderate PTSS severity according to the Child and Adolescents Trauma Screen 2 (CATS-2).
* Caregivers must have sufficient command of the German language.
* The children and adolescents do not have any physical impairment due to injuries or somatic illnesses (self-assessment).
* The children and adolescents are not acute suicidal. The responsible psychotherapists or supervisors of the "Schlupfhuus" will provide information about it.

For clinical experts:

* Clinician or researcher specialized in trauma and PTSD in children and adolescents.
* Clinical experts must have sufficient command of the English language.

Exclusion Criteria:

* For children and adolescent participants:

  * Children and Adolescents who have not experienced at least one PTE according to the DSM-5 definition of a traumatic event.
  * The PTE(s) occurred before the fourth birthday.
  * The PTE(s) occurred less than 1 month ago.
  * Children and adolescents that are younger than 7 years old and older than 18 years old.
  * Children and adolescents that are neither in trauma-focused therapy at the time of recruitment nor meet the CATS-2 score for moderate PTSS severity or higher.
  * Children and adolescents that do not have sufficient command of the German language.
  * Children and adolescents that have physical impairment due to injuries or somatic illnesses (self-assessment).
  * Children and adolescents that are acute suicidal. The responsible psychotherapists or supervisors of the "Schlupfhuus" will provide information about it.

For caregivers:

* Caregivers of children or adolescents who have not experienced at least one PTE according to the DSM-5 definition of a traumatic event.
* The PTE(s) occurred less than 1 month ago.
* The child or adolescent is younger than 1 year old or older than 18 years old.
* The child or adolescent is neither in trauma-focused therapy at the time of recruitment nor meets the CATS-2 score for moderate PTSS severity or higher.
* Caregivers that do not have sufficient command of the German language.
* Children and adolescents that have physical impairment due to injuries or somatic illnesses (self-assessment).
* Children and adolescents that are acute suicidal. The responsible psychotherapists or supervisors of the "Schlupfhuus" will provide information about it.

For clinical experts:

* Clinical experts that don't work as clinician or as researcher specialized in trauma and PTSD in children and adolescents.
* Clinical experts that do not have sufficient command of the English language.

All the participants' informed consent must be obtained before any data is collected.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Children and adolescents (7-18years old) who experienced at least one traumatic event.
  2. Caregivers of children and adolescents (1-18 years old) who experienced at least one traumatic event.
  3. Clinical experts
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
A set of relevant domains and corresponding difficulties within domains of functional impairment in trauma-exposed children and adolescents, identified in focus groups. | Oct23-Nov23
  Relevant domains of PTSD-related functional impairment in trauma-exposed children and adolescents will be identified via focus groups. Trauma-exposed children and adolescents and caregivers will participate in small focus groups.
A set of relevant domains and corresponding difficulties within domains of functional impairment in trauma-exposed children and adolescents, identified in a Delphi survey. | Nov23-Feb24
  Based on the results of the focus group discussions, relevant domains of PTSD-related functional impairment in trauma-exposed children and adolescents will be identified via Delphi survey. Trauma-exposed children and adolescents, caregivers and clinical experts will participate. Due to the exploratory design, no pre-existig scale will be used. Participants will be asked to assess the previously identified areas of PTSD-related functional impairment in children and adolescents based on their importance. For each previously identified domain, a 5-point Likert scale will be used to indicate how important it is to include that domain in the questionnaire we are developing.The scale ranges from (1) not important to (5) very important. High scores indicate that it is important to include a specific domain in the questionnaire. If the importance of a domain is rated above 1, the importance of specific difficulties within that domain will then be assessed on the same 5-point Likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University-Children's Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No